CLINICAL TRIAL: NCT02501096
Title: A Multicenter, Open-Label Phase 1b/2 Trial of Lenvatinib (E7080) Plus Pembrolizumab in Subjects With Selected Solid Tumors
Brief Title: A Trial of Lenvatinib (E7080) Plus Pembrolizumab in Participants With Selected Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-111; 2017-000300-26 (EudraCT Number)
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-06

CONDITIONS: Tumors
Keywords: Lenvatinib; Lenvima; E7080; Phase 1b/2; Pembrolizumab; Keytruda; Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenvatinib + Pembrolizumab (Experimental): Participants with one of the tumors: non-small cell lung cancer, renal cell carcinoma, endometrial cancer, urothelial cancer, squamous cell carcinoma of the head and neck, melanoma or leiomyosarcoma.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be administered with water orally once a day (with or without food) continuously in 21-day treatment cycle.
  Other Names: Lenvima; E7080
Drug: Pembrolizumab — Pembrolizumab will be administered as a dose of 200 mg Q3W, IV in 21-day treatment cycle.
  Other Names: Keytruda; MK-3475

SUMMARY:
This is an open-label Phase 1b/2 trial of lenvatinib (E7080) plus pembrolizumab in participants with selected solid tumors. Phase 1b will determine and confirm the maximum tolerated dose (MTD) for lenvatinib in combination with 200 milligrams (mg) (intravenous [IV], every 3 weeks [Q3W]) pembrolizumab in participants with selected solid tumors (i.e. non-small cell lung cancer, renal cell carcinoma, endometrial carcinoma, urothelial carcinoma, squamous cell carcinoma of the head and neck, melanoma or leiomyosarcoma). Phase 2 (Expansion) will evaluate the safety and efficacy of the combination in 7 cohorts at the MTD from Phase 1b (lenvatinib 20 mg/day orally + pembrolizumab 200 mg Q3W, IV).

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1b: Histologically and/or cytologically confirmed metastatic selected solid tumor types that have progressed after treatment with approved therapies or for which there are no standard effective therapies available. If nivolumab or pembrolizumab is an approved therapy for the participant's tumor type, but the participant has not been treated with it, the Investigator may enroll the participant in this study.

   Phase 2: Histologically and/or cytologically confirmed metastatic selected solid tumor types with 0-2 prior lines of systemic therapy. If previously treated, participant has progressed after previous treatment. For the non-small cell lung cancer (NSCLC) and melanoma cohorts, participants must have progressed on or after prior treatment with one anti-programmed cell death protein 1 (anti-PD-1), anti-PD-1 ligand 1 (anti-PD-L1), or anti-PD-1 ligand 2 (anti-PD-L2) agent. For the renal cell carcinoma (RCC) cohort, participants must have progressed on treatment with an anti- programmed death receptor-1 /programmed death receptor-ligand 1 monoclonal antibody (anti-PD-1/PD-L1 mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies, the regimen with an anti-PD-1/PD-L1 mAb must be the most recent therapy. Selected tumor types of both phases: NSCLC, predominantly clear cell renal cell carcinoma, endometrial carcinoma, urothelial carcinoma, squamous cell carcinoma of the head and neck, or melanoma (excluding uveal melanoma)
2. Life expectancy of 12 weeks or more
3. Phase 2: Measurable disease meeting the following criteria:

   1. At least 1 lesion of greater than or equal to 10 mm in the longest diameter for a non-lymph node or greater than or equal to 15 mm in the short-axis diameter for a lymph node that is serially measurable according to irRECIST (immune-related Response Evaluation Criteria in Solid Tumors) using computerized tomography/magnetic resonance imaging (CT/MRI)
   2. Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radiofrequency (RF) ablation must show subsequent evidence of substantial size increase to be deemed a target lesion
4. Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
5. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than or equal to 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the Cycle 1 Day 1
6. Adequate renal function defined as creatinine less than or equal to 1.5*ULN (upper limit of normal) or calculated creatinine clearance greater than or equal to 40 mL/min per the Cockcroft and Gault formula with creatinine levels greater than 1.5*ULN
7. Adequate bone marrow function:

   1. Absolute neutrophil count (ANC) greater than or equal to 1500/mm3 (greater than or equal to 1.5 X 103/uL)
   2. Platelets greater than or equal to 100,000/mm3 (greater than or equal to 100 X 109/L)
   3. Hemoglobin greater than or equal to 9.0 g/dL
8. Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) less than or equal to 1.5
9. Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the ULN and alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3*ULN (in the case of liver metastases less than or equal to 5*ULN). In case ALP is greater than 3 X ULN (in the absence of liver metastases) or greater than 5 X ULN (in the presence of liver metastases) AND the participant also is known to have bone metastases, the liver specific ALP must be separated from the total and used to assess the liver function instead of the total ALP
10. Males or females age greater than or equal to 18 years at the time of informed consent
11. Participants with known brain metastases will be eligible if they have completed the primary brain therapy (such as whole brain radiotherapy, stereotactic radiosurgery or complete surgical resection) and if they have remained clinically stable, asymptomatic and off of steroids for at least 28 days before starting study treatment.
12. All females must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta-human chorionic gonadotropin [β-hCG]) at the Screening Visit and the Baseline Visit. A pregnancy test needs to be performed within 72 hours of the first dose of study drug. Females of childbearing potential must agree to use a highly effective method of contraception for the entire study period and for 120 days after study discontinuation, ie

    * total abstinence (if it is their preferred and usual lifestyle)
    * an intrauterine device (IUD) or hormone-releasing system (IUS)
    * a contraceptive implant
    * an oral contraceptive** (with additional barrier method) OR
    * have a vasectomized partner with confirmed azoospermia.

    NOTES:
    * All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
    * Must be on a stable dose of the same oral hormonal contraceptive product for at least 4 weeks before dosing with study drug and for the duration of the study
13. Male participants who are partners of women of childbearing potential must use a condom + spermicide and their female partners if of childbearing potential must use a highly effective method of contraception (see methods described in Inclusion Criterion #12) beginning at least 1 menstrual cycle prior to starting study drug(s), throughout the entire study period, and for 120 days after the last dose of study drug, unless the male participants are totally sexually abstinent or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile.
14. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol
15. Archival tumor tissue or a newly obtained biopsy must be available prior to the first dose of study drug for biomarker analysis. In the case archival tissue cannot be provided, participants with inaccessible tumors for biopsy specimens can be enrolled without a biopsy upon consultation and agreement by the sponsor Note: In case of submitting unstained cut slides, freshly cut slides should be submitted to the testing laboratory within 14 days from when the slides are cut.

Exclusion Criteria:

1. Prior anticancer treatment within 28 days (or 5 times the half-life time, whichever is shorter) or any investigational agent within 30 days prior to the first dose of study drugs. All acute toxicities related to prior treatments must be resolved to Grade less than or equal to 1
2. Participants must have recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy
3. Participants having greater than 1+ proteinuria on urinalysis will undergo 24-h urine collection for quantitative assessment of proteinuria. Participants with urine protein greater than or equal to 1 g/24-hour will be ineligible.
4. Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib
5. New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months
6. Prolongation of corrected QT (QTc) interval to greater than 480 msec
7. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug
8. Active infection (any infection requiring systemic treatment)
9. Participant is known to be positive for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
10. Serious nonhealing wound, ulcer, or bone fracture
11. Known intolerance to either of the study drugs (or any of the excipients)
12. History of organ allograft (Participant has had an allogenic tissue/solid organ transplant)
13. Biologic response modifiers (eg, granulocyte colony-stimulating factor) within 4 weeks before study entry. Chronic erythropoietin therapy is permitted provided that no dose adjustments were made within 2 months before first dose of study treatment
14. Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial
15. Females who are pregnant or breastfeeding
16. Excluding the primary tumor leading to enrollment in this study, any other active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the bladder or cervix) within the past 24 months
17. Prior treatment with lenvatinib or any PD-1, anti-PD-L1, or anti-PD-L2 agent, excluding melanoma and NSCLC where prior treatment with one PD-1, anti-PD-L1, or anti-PD-L2 agent is allowed, and excluding RCC where prior treatment with one regimen containing an anti-PD-1/PD-L1 mAb is required.
18. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids (up to 7.5mg/d of prednisone or equivalent) may be approved after consultation with the sponsor.
19. No active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
20. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
21. Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (50):
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Arizona Oncology Associates, Oro Valley, Arizona
  - Arizona Oncology Associates, PC - HOPE, Site #1, Tucson, Arizona
  - Arizona Oncology Associates, PC - HOPE, Site #2, Tucson, Arizona
  - Arizona Oncology Associates, PC - HOPE, Site #3, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Site #1, Denver, Colorado
  - Rocky Mountain Cancer Centers, Site #2, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Centers, Parker, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Baptist Health Medical Group Oncology, LLC, Site #1, Miami, Florida
  - Baptist Health Medical Group Oncology, LLC, Site #2, Miami, Florida
  - Baptist Health Medical Group Oncology, LLC, Site #3, Miami, Florida
  - Boca Raton Clinical Research Medical Center, Plantation, Florida
  - Piedmont Cancer Institue, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mass General Hospital, Boston, Massachusetts
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada, Site #1, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Site #2, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Site #3, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Site #1, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Site #2, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Site #3, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Site #4, Las Vegas, Nevada
  - New York Hematology Oncology (US Onc), Albany, New York
  - Memorial Sloan Kettering at Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Oncology-Bedford, Bedford, Texas
  - Texas Oncology (US Onc), Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Texas Oncology-Fort Worth, Site #1, Fort Worth, Texas
  - Texas Oncology-Grapevine, Grapevine, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Texas Oncology-Waco, Site #1, Waco, Texas
  - Texas Oncology-Waco, Site #2, Waco, Texas
- Norway (5):
  - Haukeland Univerity Hospital, Bergen
  - Sørlandet Hospital, Kristiansand
  - Akershus Universitetssykehus HF, Lørenskog
  - Oslo Univerity Hospital, Oslo
  - Sykehuset Østfold, Sarpsborg
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario De Fuenlabrada, Fuenlabrada
  - Hospital La Paz, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - MD Anderson Cancer Center Madrid - España, Madrid
  - Parc Taulí Sabadell, Sabadell
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitari i Politécnic La Fe., Valencia

REFERENCES:
- [Derived] Makker V, Taylor MH, Aghajanian C, Cohn AL, Brose MS, Simone CD, Cao ZA, Suttner L, Loboda A, Cristescu R, Jelinic P, Orlowski R, Dutta L, Matsui J, Dutcus CE, Minoshima Y, Messing MJ. Evaluation of potential biomarkers for lenvatinib plus pembrolizumab among patients with advanced endometrial cancer: results from Study 111/KEYNOTE-146. J Immunother Cancer. 2024 Jan 19;12(1):e007929. doi: 10.1136/jitc-2023-007929. PMID 38242717
- [Derived] Makker V, Aghajanian C, Cohn AL, Romeo M, Bratos R, Brose MS, Messing M, Dutta L, Dutcus CE, Huang J, Schmidt EV, Orlowski R, Taylor MH. A Phase Ib/II Study of Lenvatinib and Pembrolizumab in Advanced Endometrial Carcinoma (Study 111/KEYNOTE-146): Long-Term Efficacy and Safety Update. J Clin Oncol. 2023 Feb 10;41(5):974-979. doi: 10.1200/JCO.22.01021. Epub 2023 Jan 6. PMID 36608305
- [Derived] Lee CH, Shah AY, Rasco D, Rao A, Taylor MH, Di Simone C, Hsieh JJ, Pinto A, Shaffer DR, Girones Sarrio R, Cohn AL, Vogelzang NJ, Bilen MA, Gunnestad Ribe S, Goksel M, Tennoe OK, Richards D, Sweis RF, Courtright J, Heinrich D, Jain S, Wu J, Schmidt EV, Perini RF, Kubiak P, Okpara CE, Smith AD, Motzer RJ. Lenvatinib plus pembrolizumab in patients with either treatment-naive or previously treated metastatic renal cell carcinoma (Study 111/KEYNOTE-146): a phase 1b/2 study. Lancet Oncol. 2021 Jul;22(7):946-958. doi: 10.1016/S1470-2045(21)00241-2. Epub 2021 Jun 15. PMID 34143969
- [Derived] Lee CH, DiNatale RG, Chowell D, Krishna C, Makarov V, Valero C, Vuong L, Lee M, Weiss K, Hoen D, Morris L, Reznik E, Murray S, Kotecha R, Voss MH, Carlo MI, Feldman D, Sachdev P, Adachi Y, Minoshima Y, Matsui J, Funahashi Y, Nomoto K, Hakimi AA, Motzer RJ, Chan TA. High Response Rate and Durability Driven by HLA Genetic Diversity in Patients with Kidney Cancer Treated with Lenvatinib and Pembrolizumab. Mol Cancer Res. 2021 Sep;19(9):1510-1521. doi: 10.1158/1541-7786.MCR-21-0053. Epub 2021 May 26. PMID 34039647
- [Derived] Makker V, Taylor MH, Aghajanian C, Oaknin A, Mier J, Cohn AL, Romeo M, Bratos R, Brose MS, DiSimone C, Messing M, Stepan DE, Dutcus CE, Wu J, Schmidt EV, Orlowski R, Sachdev P, Shumaker R, Casado Herraez A. Lenvatinib Plus Pembrolizumab in Patients With Advanced Endometrial Cancer. J Clin Oncol. 2020 Sep 10;38(26):2981-2992. doi: 10.1200/JCO.19.02627. Epub 2020 Mar 13. PMID 32167863
- [Derived] Taylor MH, Lee CH, Makker V, Rasco D, Dutcus CE, Wu J, Stepan DE, Shumaker RC, Motzer RJ. Phase IB/II Trial of Lenvatinib Plus Pembrolizumab in Patients With Advanced Renal Cell Carcinoma, Endometrial Cancer, and Other Selected Advanced Solid Tumors. J Clin Oncol. 2020 Apr 10;38(11):1154-1163. doi: 10.1200/JCO.19.01598. Epub 2020 Jan 21. PMID 31961766
- [Derived] Makker V, Rasco D, Vogelzang NJ, Brose MS, Cohn AL, Mier J, Di Simone C, Hyman DM, Stepan DE, Dutcus CE, Schmidt EV, Guo M, Sachdev P, Shumaker R, Aghajanian C, Taylor M. Lenvatinib plus pembrolizumab in patients with advanced endometrial cancer: an interim analysis of a multicentre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2019 May;20(5):711-718. doi: 10.1016/S1470-2045(19)30020-8. Epub 2019 Mar 25. PMID 30922731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 62 investigative sites in the United States, Spain and Norway from 22 July 2015 to 11 July 2022.
Pre-assignment Details: Total of 454 participants were screened, of which 357 were enrolled/treated. A total of 13 participants were enrolled in Phase 1b, of which 3 participants received lenvatinib 24 mg/day+pembrolizumab 200 mg and 10 participants received lenvatinib 20 mg/day+pembrolizumab 200 mg while in Phase 2, 344 participants received lenvatinib 20 mg/day+pembrolizumab 200 mg. As planned,Phase 1b/2 data for participants who received lenvatinib 20 mg/day+pembrolizumab 200 mg was combined and presented together.
Groups:
- Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC: Participants with Renal Cell Carcinoma (RCC) received lenvatinib 24 milligram per day (mg/day), capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, once every three weeks (Q3W) on Day 1 of each cycle (cycle length=21 days) until disease progression (PD), development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC: Participant with Non-small Cell Lung Cancer (NSCLC) received lenvatinib 24 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC: Participants with Endometrial Carcinoma (EC) received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC: Participants with RCC received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma: Participants with Melanoma received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC: Participants with NSCLC received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC: Participants with Squamous Cell Carcinoma of Head and Neck (HNSCC) received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC: Participants with Urothelial Carcinoma (UC) received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma: Participant with Leiomyosarcoma received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
Period: Overall Study
Arm/Group | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Started | 2 | 1 | 124 | 145 | 21 | 21 | 22 | 20 | 1
Phase 1b Participants Who Received, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg. | 0 | 0 | 2 | 6 | 1 | 1 | 0 | 0 | 0
Phase 2 Participants Who Received, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg | 0 | 0 | 122 | 139 | 20 | 20 | 22 | 20 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 1 | 124 | 145 | 21 | 21 | 22 | 20 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 7 | 13 | 2 | 2 | 2 | 3 | 0
Not completed — Survival follow-up discontinued by sponsor | 0 | 0 | 29 | 58 | 3 | 2 | 2 | 1 | 0
Not completed — Death | 1 | 1 | 88 | 74 | 15 | 16 | 15 | 16 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least one dose of study drug.
Groups:
- Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC: Participants with RCC received lenvatinib 24 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC: Participant with NSCLC received lenvatinib 24 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC: Participants with EC received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC: Participants with HNSCC received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC: Participants with UC received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Total: Total of all reporting groups
Arm/Group | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma | Total
Number analyzed (Participants) | 2 | 1 | 124 | 145 | 21 | 21 | 22 | 20 | 1 | 357
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 0 | 0 | 47 | 88 | 16 | 9 | 9 | 4 | 1 | 174
  >=65 years | 2 | 1 | 77 | 57 | 5 | 12 | 13 | 16 | 0 | 183
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 124 | 32 | 4 | 10 | 4 | 6 | 1 | 182
  Male | 2 | 0 | 0 | 113 | 17 | 11 | 18 | 14 | 0 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 17 | 2 | 0 | 1 | 2 | 0 | 26
  Not Hispanic or Latino | 1 | 1 | 121 | 128 | 19 | 21 | 21 | 18 | 1 | 331
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 7 | 6 | 0 | 3 | 2 | 0 | 1 | 19
  White | 2 | 1 | 108 | 125 | 19 | 18 | 20 | 19 | 0 | 312
  More than one race | 0 | 0 | 2 | 8 | 1 | 0 | 0 | 1 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Lenvatinib
Description: MTD was confirmed if no more than 3 participants experience dose-limiting toxicities(DLTs)during first 3 weeks (Cycle 1) of treatment.If MTD was not confirmed at dose level,then enrollment was proceeded to next lower dose level.Sponsor and investigators reviewed all participants' safety;clinical data to jointly determine RP2D of combination of treatment.DLT may be any of following: hematological/nonhematological toxicities considered to be at least possibly related to Lenvatinib/pembrolizumab occurring during Cycle 1;Failure to administer greater than or equal to (>=) 75 percent (%) of planned dosage of lenvatinib as result of treatment-related toxicity during Cycle 1;Who discontinue treatment due to treatment-related toxicity.Greater than 2 week delay in starting Cycle 2 because of treatment-related toxicity,even if toxicity does not meet DLT criteria.Toxicity was evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03(NCI CTCAE v 4.03).
Time Frame: Cycle 1 (21 days)
Population: The MTD analysis set included all participants who completed Cycle 1 of treatment in Phase 1b or discontinued early due to DLT.
Measure: Number; unit: milligram (mg)
Groups:
- Phase 1b: All Participants: All participants with selected solid tumors (RCC, EC, NSCLC and Melanoma) received lenvatinib 24 or 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
Arm/Group | Phase 1b: All Participants
Number analyzed (Participants) | 13
milligram (mg)
  MTD | 20
  RP2D | 20

2. Primary Outcome: Phase 1b: Number of Participants With Dose Limiting Toxicities (DLTs) of Lenvatinib
Description: A DLT was defined as any of the following: any of the hematological or nonhematological toxicities considered to be at least possibly related to lenvatinib and/or pembrolizumab occurring during Cycle 1. Failure to administer >=75% of the planned dosage of lenvatinib as a result of treatment-related toxicity during Cycle 1. Participants who discontinue treatment due to treatment-related toxicity. Greater than 2 week delay in starting Cycle 2 because of a treatment-related toxicity, even if the toxicity does not meet DLT criteria. Toxicity was evaluated as per NCI CTCAE v 4.03.
Time Frame: Cycle 1 (21 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg: NSCLC: Participant with NSCLC received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg: RCC: Participants with RCC received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg: EC: Participant with EC received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
- Phase 1b, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg: Melanoma: Participant with Melanoma received lenvatinib 20 mg/day, capsules, orally, once daily in combination with pembrolizumab 200 mg, intravenous, infusion, Q3W on Day 1 of each cycle (cycle length=21 days) until PD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor.
Arm/Group | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC | Phase 1b, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg: NSCLC | Phase 1b, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg: RCC | Phase 1b, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg: EC | Phase 1b, Lenvatinib 20 mg/Day + Pembrolizumab 200 mg: Melanoma
Number analyzed (Participants) | 2 | 1 | 1 | 6 | 2 | 1
Participants | 1 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Objective Response Rate (ORR) Based on Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) Version 1.1 at Week 24
Description: ORR was defined as the percentage of participants whose best overall response (BOR) was immune related complete response (irCR) or immune related partial response (irPR) based on investigator assessment according to irRECIST version 1.1. irCR was defined as disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). irPR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Week 24
Population: The full analysis set (FAS) included all participants who entered the study treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 124 | 145 | 21 | 21 | 22 | 20 | 1
percentage of participants | 39.5 [30.9 to 48.7] | 56.6 [48.1 to 64.8] | 47.6 [25.7 to 70.2] | 23.8 [8.2 to 47.2] | 31.8 [13.9 to 54.9] | 25.0 [8.7 to 49.1] | 0 [NA to NA] — Here, 95% CI could not be estimated as insufficient number of participants were available for analysis in this arm.

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: TEAE: adverse event (AE) emerged during treatment, having been absent at pretreatment or reemerged during treatment, present at pretreatment but stopped before treatment or worsened in severity during treatment relative to pretreatment state, when AE is continuous. AE: any untoward medical occurrence in participant administered an investigational product. TEAEs were based on participants laboratory tests, regular measurement of vital signs, echocardiograms/multigated acquisition scans to assess left ventricular ejection fraction and electrocardiograms parameter values. TESAE: any untoward medical occurrence that at any dose: resulted in death; life threatening condition; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; a congenital anomaly/birth defect or was medically important due to reasons other than above criteria.
Time Frame: From date of first dose up to 30 days after the last dose of study drugs (Up to 74 months)
Population: The safety analysis set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 2 | 1 | 124 | 145 | 21 | 21 | 22 | 20 | 1
Participants
  TEAEs | 2 | 1 | 124 | 145 | 21 | 21 | 22 | 20 | 1
  TESAEs | 1 | 1 | 73 | 81 | 12 | 15 | 12 | 17 | 0

5. Secondary Outcome: Objective Response Rate (ORR) Based on irRECIST Version 1.1
Description: ORR was defined as the percentage of participants whose BOR was irCR or irPR according to irRECIST version 1.1. irCR was defined as disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. irPR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first dose of study drug administration until immune related (irPD), development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor (up to 73 months)
Population: The FAS included all participants who entered the study treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 124 | 145 | 21 | 21 | 22 | 20 | 1
percentage of participants | 40.3 [31.6 to 49.5] | 63.4 [55.1 to 71.3] | 47.6 [25.7 to 70.2] | 23.8 [8.2 to 47.2] | 40.9 [20.7 to 63.6] | 25.0 [8.7 to 49.1] | NA [NA to NA] — Here, number and 95% CI could not be estimated as insufficient number of participants were available for analysis in this arm.

6. Secondary Outcome: Progression-free Survival (PFS) Based on irRECIST Version 1.1
Description: PFS was defined as the time from the first dose date to the date of irPD or date of death (whichever occurred first) according to irRECIST version 1.1. irPD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions was also considered progression).
Time Frame: From date of first dose of study drug administration to date of irPD or date of death, whichever occurred first (up to 73 months)
Population: The FAS included all participants who entered the study treatment period.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 124 | 145 | 21 | 21 | 22 | 20 | 1
months | 7.5 [5.3 to 9.7] | 14.1 [11.6 to 18.4] | 5.5 [2.6 to 15.8] | 5.4 [2.3 to 7.4] | 4.4 [4.0 to 9.8] | 5.4 [1.3 to 42.3] | 1.35 [NA to NA] — Here, 95% CI could not be estimated as insufficient number of participants were available for analysis in this arm.

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose date to the date of death from any cause.
Time Frame: From the first dose until death from any cause, up to 73 months
Population: The FAS included all participants who entered the study treatment period.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 124 | 145 | 21 | 21 | 22 | 20 | 1
months | 19.9 [16.2 to 25.9] | 32.2 [29.8 to 55.8] | 25.4 [8.6 to 39.5] | 11.4 [3.6 to 23.3] | 16.2 [8.6 to 31.8] | 6.1 [2.4 to 30.1] | 16.56 [NA to NA] — Here, 95% CI could not be estimated as insufficient number of participants were available for analysis in this arm.

8. Secondary Outcome: Disease Control Rate (DCR) Based on irRECIST Version 1.1
Description: DCR: percentage of participants with a confirmed irCR, irPR, or ir-stable disease (SD) (duration of irSD greater than or equal to [>=] 5 weeks). DCR was assessed on irRECIST v1.1. irCR: disappearance of all target lesions. All pathological lymph nodes (whether target or non-target) must have reduction in their short axis to <10 mm. irPR: at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference baseline sum of longest diameter. irSD: neither sufficient shrinkage to qualify for irPR nor sufficient increase to qualify for irPD, taking as reference smallest sum diameters while on study. irPD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study).
Time Frame: From first dose of the study drug until irPD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor (up to 73 months)
Population: The FAS included all participants who entered the study treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 124 | 145 | 21 | 21 | 22 | 20 | 1
percentage of participants | 84.7 [77.1 to 90.5] | 93.8 [88.5 to 97.1] | 81.0 [58.1 to 94.6] | 76.2 [52.8 to 91.8] | 90.9 [70.8 to 98.9] | 70.0 [45.7 to 88.1] | NA [NA to NA] — Here, Number and 95% CI could not be estimated as insufficient number of participants were available for analysis in this arm.

9. Secondary Outcome: Clinical Benefit Rate (CBR) Based on irRECIST Version 1.1
Description: CBR was defined as the percentage of participants with BOR of irCR or irPR or irdurable stable disease (irdSD) (duration of irSD >=23 weeks) [irCR + irPR + irdSD] based on irRECIST v1.1. irCR: disappearance of all target lesions. All pathological lymph nodes (whether target or non-target) must have reduction in their short axis to <10 mm. irPR: at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference baseline sum of longest diameter. irSD: neither sufficient shrinkage to qualify for irPR nor sufficient increase to qualify for irPD, taking as reference smallest sum diameters while on study. irPD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study).
Time Frame: From first dose date until irPD, development of unacceptable toxicity, participant choice, withdrawal of consent, lost to follow up or discontinuation of this study by the sponsor (up to 73 months)
Population: The FAS included all participants who entered the study treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 124 | 145 | 21 | 21 | 22 | 20 | 1
percentage of participants | 58.9 [49.7 to 67.6] | 80.0 [72.6 to 86.2] | 61.9 [38.4 to 81.9] | 57.1 [34.0 to 78.2] | 45.5 [24.4 to 67.8] | 40.0 [19.1 to 63.9] | NA [NA to NA] — Here, Number and 95% CI could not be estimated as insufficient number of participants were available for analysis in this arm.

10. Secondary Outcome: Durable Stable Disease Rate (DSDR) Based on irRECIST Version 1.1
Description: Durable SD rate is defined as the percentage of participants whose observed BOR is irSD and the duration of irSD is >=23 weeks based on irRECIST v1.1.
Time Frame: as for outcome 9
Population: The FAS included all participants who entered the study treatment period. As planned, data for this outcome measure dSD rate (where SD>=23 weeks) was not analyzed and collected separately but was included and analyzed in outcome measure CBR (irCR+irPR+[irSD duration >=23 weeks]).
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Duration of Objective Response (DOR) Based on irRECIST Version 1.1
Description: DOR: time from date of first observation of response (irPR or irCR) to date of the first observation of progression based on irRECIST 1.1, or date of death, whatever the cause. irCR: disappearance of all target and non-target lesions. All pathological (whether target or non-target) must have reduction in their short axis <10 mm. irPR: at least 30% decrease in sum of diameter (SOD) of target lesions, taking as reference baseline sum diameters. irPD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in SOD of target lesions, taking as reference smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: First documentation of irCR or irPR until first documentation of progression or death (up to 73 months)
Population: The FAS included all participants who entered the study treatment period. Here "overall number of participants analyzed, N" signifies participants who had irCR or irPR. Here, "N" for Phase1b and 2, Lenvatinib 20 mg/day + Pembrolizumab 200 mg: Leiomyosarcoma was zero as there were no events of irCR or irPR in this arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 50 | 92 | 10 | 5 | 9 | 5 | 0
months | NA [8.5 to NA] — Median and Upper limit of 95% CI could not be estimated because high number of participants in this arm were censored from the analyses. | 16.6 [9.7 to 18.4] | 12.5 [2.7 to 28.6] | 14.5 [2.4 to NA] — Here, Upper limit of 95% CI could not be estimated as insufficient number of participants were available for analysis in this arm. | 7.1 [2.2 to 16.8] | 41.0 [4.6 to NA] — Here, Upper limit of 95% CI could not be estimated as insufficient number of participants were available for analysis in this arm. |

12. Secondary Outcome: Phase 1b: Plasma Concentrations of Lenvatinib
Description: Observed plasma concentration of Lenvatinib was reported here quantified by liquid chromatography with tandem mass spectrometry (LCMS/MS) method.
Time Frame: Cycle 1 Day 1: 0.5-4 hours and 6-10 hours post dose; Cycle 1 Day 15: predose, 0.5-4 hours and 6-10 hours post dose, Cycle 2 Day 1: predose, 2-12 hour postdose and Cycles 3,4,5,6 Day 1 predose (Cycle length =21 days)
Population: The Pharmacokinetic (PK) analysis set included all participants who had received at least 1 dose of lenvatinib and had evaluable concentration data. Here number analyzed "n" signifies number of participants who were evaluable for given time points.
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC
Number analyzed (Participants) | 2 | 1
microgram per liter (mcg/L)
  Cycle 1 Day 1: 0.5-4 hour | 102.5 (136.44) | 198.0 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 1 Day 1: 6-10 hour: number analyzed (Participants) | 2 | 0
  Cycle 1 Day 1: 6-10 hour | 210.5 (65.76) |
  Cycle 1 Day 15: Predose: number analyzed (Participants) | 1 | 1
  Cycle 1 Day 15: Predose | 53.9 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 1.8 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 1 Day 15: 0.5-4 hour: number analyzed (Participants) | 1 | 1
  Cycle 1 Day 15: 0.5-4 hour | 78.4 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 2.6 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 1 Day 15: 6-10 hour: number analyzed (Participants) | 1 | 1
  Cycle 1 Day 15: 6-10 hour | 366.0 (NA) — Standard deviation could not be calculated because only one participant was available for analysis. | 424.0 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 2 Day 1: Predose | 35.4 (13.08) | 364.0 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 2 Day 1: 2-12 hour | 491.0 (247.49) | 374.0 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 3 Day 1: Predose | 23.3 (31.92) | 118.0 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 4 Day 1: Predose | 28.0 (13.93) | 176.0 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 5 Day 1: Predose | 19.9 (14.91) | 2.5 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 6 Day 1: Predose | 44.4 (42.64) | 210.0 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.

13. Secondary Outcome: Plasma Concentrations of Lenvatinib
Description: Observed plasma concentration of Lenvatinib was reported here quantified by LCMS/MS method.
Time Frame: Cycle 1 Day 1: 0.5-4 hours and 6-10 hours post dose; Cycle 1 Day 15: predose, 0.5-4 hours and 6-10 hours post dose, Cycle 2 Day 1: predose, 2-12 hour postdose and Cycles 3,4,5,6 Day 1 predose (Cycle length =21 days):
Population: The PK analysis set included all participants who had received at least 1 dose of lenvatinib and had evaluable concentration data. Here, overall number of participants analyzed, N signifies participants who were evaluable for this outcome measure and number analyzed "n" signifies number participants who were evaluable for given time points.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
Number analyzed (Participants) | 122 | 138 | 20 | 20 | 22 | 20 | 1
mcg/L
  Cycle 1 Day 1:0.5-4 hour: number analyzed (Participants) | 122 | 138 | 20 | 20 | 22 | 20 | 0
  Cycle 1 Day 1:0.5-4 hour | 82.2 (145.44) | 35.5 (78.13) | 24.0 (33.59) | 79.9 (118.94) | 41.8 (100.34) | 123.8 (169.05) |
  Cycle 1 Day 1:6-10 hour: number analyzed (Participants) | 116 | 111 | 18 | 16 | 19 | 16 | 1
  Cycle 1 Day 1:6-10 hour | 231.7 (109.67) | 190.8 (96.25) | 154.3 (69.56) | 224.1 (109.95) | 169.7 (95.78) | 214.2 (86.51) | 116 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 1 Day 15:Predose: number analyzed (Participants) | 103 | 125 | 16 | 13 | 16 | 14 | 1
  Cycle 1 Day 15:Predose | 66.6 (36.56) | 67.2 (80.70) | 52.1 (61.70) | 62.9 (87.36) | 60.9 (46.38) | 61.1 (69.54) | 52.2 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 1 Day 15:0.5-4 hour: number analyzed (Participants) | 103 | 117 | 18 | 13 | 17 | 15 | 1
  Cycle 1 Day 15:0.5-4 hour | 129.3 (109.72) | 122.4 (114.62) | 93.1 (117.35) | 275.3 (305.30) | 142.8 (149.90) | 153.9 (135.79) | 45.9 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 1 Day 15:6-10 hour: number analyzed (Participants) | 99 | 104 | 17 | 13 | 15 | 15 | 1
  Cycle 1 Day 15:6-10 hour | 271.3 (103.60) | 206.3 (97.29) | 241.8 (241.52) | 266.8 (146.41) | 210.6 (78.37) | 249.7 (91.65) | 161 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 2 Day 1:Predose: number analyzed (Participants) | 109 | 134 | 20 | 17 | 19 | 13 | 1
  Cycle 2 Day 1:Predose | 57.2 (60.58) | 54.6 (64.43) | 49.2 (46.63) | 51.6 (66.72) | 42.0 (48.16) | 22.3 (21.61) | 26.1 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 2 Day 1:2-12 hour: number analyzed (Participants) | 101 | 120 | 17 | 13 | 15 | 9 | 0
  Cycle 2 Day 1:2-12 hour | 199.7 (155.08) | 171.7 (119.34) | 218.6 (83.83) | 295.0 (190.80) | 166.5 (128.95) | 204.7 (174.60) |
  Cycle 3 Day 1:Predose: number analyzed (Participants) | 105 | 128 | 17 | 15 | 18 | 12 | 0
  Cycle 3 Day 1:Predose | 53.2 (59.53) | 59.0 (67.58) | 62.8 (65.77) | 99.4 (132.33) | 43.7 (50.45) | 37.9 (29.19) |
  Cycle 4 Day 1:Predose: number analyzed (Participants) | 100 | 124 | 15 | 15 | 18 | 11 | 1
  Cycle 4 Day 1:Predose | 50.7 (52.16) | 56.0 (61.56) | 65.8 (115.31) | 53.4 (81.66) | 34.3 (54.94) | 18.8 (34.33) | 61.9 (NA) — Standard deviation could not be calculated because only one participant was available for analysis.
  Cycle 5 Day 1:Predose: number analyzed (Participants) | 88 | 121 | 14 | 12 | 17 | 11 | 0
  Cycle 5 Day 1:Predose | 53.5 (56.69) | 52.1 (65.15) | 60.8 (58.38) | 71.8 (134.39) | 37.7 (42.97) | 39.0 (29.50) |
  Cycle 6 Day 1:Predose: number analyzed (Participants) | 79 | 111 | 13 | 10 | 14 | 8 | 0
  Cycle 6 Day 1:Predose | 40.6 (33.66) | 51.8 (49.19) | 114.0 (189.97) | 49.9 (68.97) | 36.9 (34.12) | 34.2 (31.86) |

ADVERSE EVENTS:
Time Frame: From date of first dose of the study drugs up to 30 days after the last dose (up to 74 months)
Description: The safety analysis set included all participants who received at least one dose of study drug.
Arm/Group | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/1 | 88/124 | 74/145 | 15/21 | 16/21 | 15/22 | 16/20 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 73/124 | 81/145 | 12/21 | 15/21 | 12/22 | 17/20 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 122/124 | 145/145 | 21/21 | 21/21 | 22/22 | 20/20 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC (N=2) | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC (N=1) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC (N=124) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC (N=145) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma (N=21) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC (N=21) | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC (N=22) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC (N=20) | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma (N=1)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 6 (8) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypobarism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (2) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (7) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 6 (7) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 8 (9) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: RCC (N=2) | Phase 1b, Lenvatinib 24 mg/Day + Pembrolizumab 200 mg: NSCLC (N=1) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: EC (N=124) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: RCC (N=145) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: Melanoma (N=21) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: NSCLC (N=21) | Phase 1b and 2,Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: HNSCC (N=22) | Phase 1b and 2, Lenvatinib 20 mg/Day+Pembrolizumab 200 mg: UC (N=20) | Phase1b and 2, Lenvatinib 20mg/Day+Pembrolizumab 200 mg: Leiomyosarcoma (N=1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 61 (77) | 60 (66) | 7 (10) | 8 (8) | 6 (7) | 8 (8) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0) | 10 (13) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 41 (50) | 43 (55) | 9 (14) | 7 (9) | 5 (5) | 5 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 1 (3) | 79 (270) | 97 (330) | 13 (23) | 12 (39) | 8 (26) | 11 (36) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 12 (13) | 21 (30) | 3 (3) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 66 (144) | 74 (132) | 13 (24) | 10 (18) | 9 (11) | 12 (19) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (4) | 1 (1) | 45 (79) | 63 (109) | 1 (1) | 5 (6) | 7 (13) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 56 (137) | 44 (84) | 9 (13) | 8 (14) | 6 (7) | 10 (12) | 1 (1)
Fatigue (General disorders) | 2 (6) | 1 (3) | 66 (159) | 95 (261) | 14 (21) | 15 (33) | 11 (25) | 12 (21) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 37 (59) | 8 (19) | 6 (8) | 3 (5) | 2 (4) | 9 (14) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 15 (28) | 18 (33) | 3 (5) | 1 (4) | 2 (5) | 3 (5) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 45 (103) | 46 (79) | 5 (13) | 7 (21) | 5 (6) | 6 (9) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 68 (135) | 70 (114) | 10 (15) | 16 (30) | 10 (14) | 10 (18) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 35 (65) | 20 (44) | 1 (1) | 4 (4) | 2 (2) | 2 (6) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 15 (21) | 21 (47) | 2 (2) | 5 (9) | 4 (10) | 4 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 49 (99) | 70 (123) | 7 (9) | 8 (16) | 4 (4) | 7 (8) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 25 (38) | 36 (47) | 3 (4) | 4 (6) | 3 (3) | 5 (5) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 28 (39) | 20 (39) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 19 (24) | 30 (38) | 3 (4) | 6 (6) | 4 (4) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 42 (62) | 44 (65) | 5 (6) | 2 (3) | 6 (8) | 4 (4) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (2) | 37 (121) | 67 (168) | 7 (13) | 8 (23) | 5 (20) | 13 (38) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 37 (62) | 59 (78) | 10 (12) | 5 (9) | 6 (6) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 9 (10) | 28 (41) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 8 (13) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 4 (5) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (2) | 75 (173) | 66 (175) | 9 (12) | 8 (25) | 8 (16) | 9 (15) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 11 (16) | 19 (31) | 2 (4) | 3 (3) | 4 (5) | 6 (7) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 9 (17) | 0 (0) | 1 (3) | 3 (4) | 1 (1) | 3 (4) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 7 (10) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 10 (10) | 1 (1) | 3 (6) | 2 (2) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 7 (7) | 6 (7) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 5 (6) | 8 (8) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 8 (11) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 38 (58) | 37 (52) | 5 (5) | 5 (6) | 1 (2) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 12 (16) | 14 (24) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 5 (5) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 22 (30) | 20 (23) | 3 (3) | 3 (4) | 1 (1) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 11 (15) | 5 (6) | 1 (1) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 15 (16) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 18 (21) | 9 (9) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 9 (9) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 11 (15) | 11 (12) | 5 (6) | 1 (1) | 6 (22) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6) | 13 (17) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 22 (70) | 6 (12) | 1 (1) | 2 (3) | 1 (1) | 4 (6) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 14 (16) | 11 (12) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 8 (8) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 29 (38) | 27 (37) | 5 (6) | 5 (12) | 3 (4) | 6 (16) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 4 (6) | 15 (18) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 13 (16) | 21 (28) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 8 (12) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 4 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 14 (17) | 9 (9) | 6 (9) | 4 (4) | 2 (2) | 2 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 13 (16) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 6 (7) | 8 (12) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 17 (37) | 18 (35) | 3 (5) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 7 (20) | 20 (67) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 14 (21) | 17 (31) | 2 (4) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 9 (12) | 7 (7) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 6 (8) | 9 (14) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 13 (26) | 29 (71) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 12 (15) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 8 (9) | 6 (11) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 20 (44) | 32 (114) | 0 (0) | 0 (0) | 0 (0) | 4 (18) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 4 (11) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 1 (6) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 5 (7) | 7 (9) | 1 (1) | 1 (3) | 2 (3) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 17 (23) | 11 (17) | 3 (3) | 4 (8) | 1 (1) | 10 (12) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 11 (13) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (10) | 11 (12) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 15 (32) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (11) | 29 (102) | 1 (1) | 1 (1) | 2 (4) | 2 (7) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (8) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 7 (13) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 19 (33) | 10 (12) | 5 (5) | 5 (8) | 1 (1) | 2 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 12 (16) | 4 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 10 (17) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 13 (18) | 17 (24) | 2 (2) | 1 (3) | 2 (3) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 13 (14) | 13 (15) | 4 (4) | 5 (6) | 1 (1) | 4 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 8 (12) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 20 (26) | 20 (31) | 2 (3) | 3 (4) | 1 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (8) | 8 (8) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 15 (20) | 28 (49) | 4 (4) | 4 (6) | 1 (1) | 4 (5) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 14 (19) | 20 (24) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 11 (12) | 10 (11) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 3 (6) | 3 (3) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 9 (10) | 11 (11) | 0 (0) | 5 (6) | 2 (2) | 2 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 5 (6) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 9 (10) | 5 (5) | 1 (2) | 3 (5) | 1 (1) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 14 (18) | 24 (29) | 4 (4) | 3 (3) | 2 (2) | 4 (7) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 7 (8) | 4 (5) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (8) | 12 (16) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 6 (7) | 11 (11) | 1 (1) | 0 (0) | 1 (4) | 1 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 33 (44) | 67 (103) | 4 (5) | 5 (8) | 7 (8) | 6 (13) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 22 (26) | 43 (68) | 3 (3) | 8 (17) | 4 (6) | 8 (11) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 13 (21) | 21 (32) | 2 (2) | 3 (4) | 1 (3) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 9 (12) | 24 (31) | 7 (7) | 3 (3) | 7 (21) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (8) | 0 (0) | 4 (5) | 1 (1) | 3 (40) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 27 (47) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 11 (12) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 11 (12) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 15 (16) | 26 (33) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 8 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 34 (80) | 46 (112) | 4 (5) | 0 (0) | 4 (7) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 19 (22) | 21 (28) | 1 (1) | 6 (13) | 2 (2) | 2 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 10 (22) | 25 (37) | 3 (3) | 3 (6) | 2 (2) | 4 (12) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 20 (36) | 25 (44) | 5 (6) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 10 (13) | 12 (13) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02501096/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT02501096/SAP_001.pdf